CLINICAL TRIAL: NCT02308111
Title: A Phase 4, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study Evaluating the Effect of Obeticholic Acid on Clinical Outcomes in Patients With Primary Biliary Cholangitis
Brief Title: Phase 4 Study of Obeticholic Acid Evaluating Clinical Outcomes in Patients With Primary Biliary Cholangitis
Acronym: COBALT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The DMC made the recommendation to not pursue further enrollment given the lack of feasibility for this post-marketing study as designed.
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 747-302
Record Dates: First submitted 2014-11-10; First posted 2014-12-04 (Estimated); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: Primary Biliary Cirrhosis; PBC; Cirrhosis; Liver
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fibrosis | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obeticholic Acid (OCA) 5 mg to 10 mg (Experimental): Obeticholic Acid (OCA) 5 mg for a minimum 3 months and then titrating up to a maximum 10 mg for the remainder of the trial (based on tolerability and CP Score).
  Interventions: Drug: Obeticholic Acid (OCA)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic Acid (OCA) — Non-cirrhotic and classified as CP Class A: 5 mg tablet of OCA once daily titrating up to a maximum of 10 mg OCA once daily based on tolerability at 3 months for the duration of the study (majority of participants).
  Cirrhotic and classified as CP Class B and C: 5 mg tablet of OCA once weekly for at least 3 months, subsequently titrating up to a maximum dose and frequency of 10 mg OCA twice weekly based on tolerability and biochemical response for the duration of the study.
  Other Names: 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
  Arms: Obeticholic Acid (OCA) 5 mg to 10 mg
Drug: Placebo — One tablet daily (or a lower frequency depending on CP score) for the remainder of the study
  Arms: Placebo

SUMMARY:
Primary Biliary Cholangitis (PBC) is a serious, life-threatening, bile acid related liver disease of unknown cause. Without treatment, it frequently progresses to liver fibrosis and eventual cirrhosis requiring liver transplantation or resulting in death. The investigational drug, Obeticholic Acid (OCA) is a modified bile acid and FXR agonist that is derived from the primary human bile acid chenodeoxycholic acid. The key mechanisms of action of OCA, including its choleretic, anti-inflammatory, and anti-fibrotic properties, underlie its hepatoprotective effects and result in attenuation of injury and improved liver function in a cholestatic liver disease such as PBC. The study will assess the effect of OCA compared to placebo, combined with stable standard care, on clinical outcomes in PBC participants.

DETAILED DESCRIPTION:
This Phase 4, double-blind, randomized, placebo-controlled, multicenter study is being undertaken at up to 170 sites internationally to evaluate the effect of OCA on clinical outcomes in 428 participants with PBC. The study will include a screening period of up to 8 weeks, requiring two clinic visits. Eligible participants will be randomly allocated (1:1) to treatment with either OCA 5 mg or matching placebo tablets, taken orally once daily for the majority of participants; dose and frequency will be modified for participants with cirrhosis and classified as Child-Pugh (CP) B or C. Randomization will be stratified by standard treatment with UDCA (yes/no) and baseline liver function. The treatment period involves clinic visits approximately every 3 months. At the 3 month visit or any study visit thereafter, if study treatment is tolerated, participants' dose should be titrated per protocol in a blinded manner eg for participants who are non-cirrhotic or classified as CP A and randomized to OCA, they should receive the maximum daily dose of 10 mg OCA, those on placebo continue to receive placebo. Subsequently, daily dosage may return to 5 mg if necessary for these participants who are non-cirrhotic or classified as CP A, but should be increased to 10 mg if possible, based on tolerability and clinical judgment. Safety and tolerability will be assessed by monitoring adverse events and vital signs, and blood and urine testing. The study is event driven and total duration will be determined by the time required to accrue approximately 127 primary endpoint events, estimated to be approximately 10 years. Participants are expected to have a minimum follow-up time of approximately 6 years.

ELIGIBILITY:
Key Inclusion Criteria:

1. Definite or probable PBC diagnosis (consistent with American Association for the Study of Liver Diseases [AASLD] and the European Association for the Study of the Liver [EASL] practice guidelines; Lindor 2009; EASL 2009), as demonstrated by the presence of ≥2 of the following 3 diagnostic factors:

   * History of elevated Alkaline phosphatase levels for at least 6 months
   * Positive antimitochondrial antibody (AMA) titer or if AMA negative or in low titer (<1:80) PBC-specific antibodies (anti-GP210 and/or anti-SP100 and/or antibodies against the major M2 components [PDC-E2, 2-oxo-glutaric acid dehydrogenase complex])
   * Liver biopsy consistent with PBC
2. A mean total bilirubin >ULN and ≤5x ULN and/or a mean ALP >3x ULN
3. Either is not taking UDCA (no UDCA dose in the past 3 months) or has been taking UDCA for at least 12 months with a stable dose for ≥3 months prior to Day 0

Exclusion Criteria:

1. History or presence of other concomitant liver diseases including:

   * Hepatitis C virus infection
   * Active Hepatitis B infection; however, subjects who have seroconverted (hepatitis B surface antigen and hepatitis B e antigen negative) may be included in this study after consultation with the medical monitor
   * Primary sclerosing cholangitis (PSC)
   * Alcoholic liver disease
   * Definite autoimmune liver disease or overlap hepatitis
   * Nonalcoholic steatohepatitis (NASH)
   * Gilbert's Syndrome
2. Presence of clinical complications of PBC or clinically significant hepatic decompensation, including:

   * History of liver transplant, current placement on a liver transplant list, or current Model of End Stage Liver Disease (MELD) score >12. Subjects who are placed on a transplant list despite a relatively early disease stage (for example per regional guidelines) may be eligible as long as they do not meet any of the other exclusion criteria
   * Cirrhosis with complications, including history (within the past 12 months) or presence of:

     * Variceal bleed
     * Uncontrolled ascites
     * Encephalopathy
     * Spontaneous bacterial peritonitis
   * Known or suspected HCC
   * Prior transjugular intrahepatic portosystemic shunt procedure
   * Hepatorenal syndrome (type I or II) or screening (Visit 1 or 2) serum creatinine >2 mg/dL (178 μmol/L)
3. Mean total bilirubin >5x ULN
4. Subjects who have undergone gastric bypass procedures (gastric lap band is acceptable) or ileal resection or plan to undergo either of these procedures
5. Other medical conditions that may diminish life expectancy, including known cancers (except carcinomas in situ or other stable, relatively benign conditions)
6. If female: plans to become pregnant, known pregnancy or a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating
7. Known history of human immunodeficiency virus infection
8. Medical conditions that may cause nonhepatic increases in ALP (eg, Paget's disease or fractures within 3 months)
9. Other clinically significant medical conditions that are not well controlled or for which medication needs are anticipated to change during the study
10. History of alcohol abuse or other substance abuse within 1 year prior to Day 0
11. Participation in another investigational product, biologic, or medical device study within 30 days prior to Screening. Participation in a previous study of OCA is allowed with 3 months washout prior to enrollment in this study
12. Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain
13. History of known or suspected clinically significant hypersensitivity to OCA or any of its components
14. UDCA naïve (unless contraindicated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2014-12-26 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Ness, MD, Study Director — Intercept Pharmaceuticals
Locations (181):
- United States (43):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California Davis, Davis Medical Center, Sacramento, California
  - Stanford University, Stanford, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Louisville, Medical Dental Complex, Louisville, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - UMass Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Southern Therapy and Advanced Research (STAR), Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Saint Louis University Gastroenterology & Hepatology, St Louis, Missouri
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Mount Sinai Beth Israel, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Texas Digestive Disease Consultants, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor Scott and White Research Institute, Fort Worth, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - UT Health The University of Texas Health Science Center at Houston, Houston, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Clinical Research Centers of America, Murray, Utah
  - McGuire DVAMC, Richmond, Virginia
  - Swedish Organ Transplant & Liver Center, Seattle, Washington
- Argentina (12):
  - Centro De Hepatología, La Plata, Buenos Aires
  - Hospital Universitario Austral, Presidente Derqui, Buenos Aires
  - Dim Clínica Privada, Ramos Mejía, Buenos Aires
  - Hospital Privado Universitario de Cordoba S.A., Córdoba, Córdoba Province
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
  - CIPREC - Centro de Investigacion y Prevencion Cardiovascular S.A., Buenos Aires
  - Hospital De Clinicas University Of Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital de Gastroenterologia Dr. Carlos Bonorino Udaondo, Buenos Aires
  - Centrol Integral de Gastroenterologia, Buenos Aires
  - Hospital Aleman, Buenos Aires
  - Hospital Britanico De Buenos Aires, Buenos Aires
- Australia (9):
  - AW Morrow Gastroenterology and Liver Centre, Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Department of Gastroenterology & Hepatology, Nepean Hospital, Kingswood, New South Wales
  - Gallipoli Medical Research Foundation, Brisbane, Queensland
  - Department of Gastroenterology and Hepatology, Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Fiona Stanley Hospital, Gastroenterology Department, Murdoch, Western Australia
- AKH, Medical University of Vienna, Vienna, Austria
- Belgium (4):
  - University Hospital Antwerp, Edegem, Antwerp
  - Uz Leuven, Leuven, Vlaams-Brabant
  - Cub Hôpital Erasme, Brussels
  - University Hospital Ghent, Ghent
- Brazil (11):
  - Gastrocentro/ Universidade Estadual de Campinas (UNICAMP), São Paulo, Campinas
  - Instituto Hospital de Base do Distrito Federal-IHBDF, Brasília, Distrito Federal Brazil
  - Hospital Sao Rafael, São Salvador, Estado de Bahia
  - Instituto Goiano de Gastroenterologia, Goiânia, Goiás
  - Cepec Huufma, São Luís, Maranhão
  - Hospital das Clinicas da Universidade Federal de Minas Gerais (UFMG), Belo Horizonte, Minas Gerais
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Universitario Professor Edgard Santos, Bahia, Salvador
  - Gastrocentro. Unidad Estadual de CAmpinas UNICAMP, Campinas, São Paulo
  - Universidade Federal do Estado do Rio de Janeiro - Hospital Universitario Gaffree e Guinle/HUGG/UNIRIO, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo-HCFMUSP, São Paulo
- St. Ivan Rilsky University Hospital, Sofia, Bulgaria
- Canada (6):
  - University of Calgary Liver Unit (Heritage Medical Research Clinic), Calgary, Alberta
  - University of Alberta, Walter C. Mackenzie Health Sciences Centre (WMC), Edmonton, Alberta
  - University Of Manitoba, Health Sciences Centre, Winnipeg, Manitoba
  - London Health Sciences Centre-University Hospital, London, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - Chum, Montreal, Quebec
- Centro De Investigaciones Clínicas Viña Del Mar, Viña del Mar, Región de Valparaíso, Chile
- Denmark (3):
  - Aarhus University Hospital Department of Hepatology and Gastroenterology, Aarhus, Aarhus C
  - Medicinsk klinik for mave, tarm-og leversygdomme, København Ø
  - Odense University Hospital Afdeling for medicinske mave-tarmsygdomme S, Odense
- Estonia (2):
  - East Tallinn Central Hospital Gastroenterology Center, Tallinn, Harju
  - Tartu University Hospital, Tartu
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Turku University Central Hospital, Gastroenterology Outpatient Clinic, Turku
- France (3):
  - Hospital Saint-Antoine, A.P.-H.P., Paris, Paris
  - CHRU Hôpital HURIEZ, Lille
  - Chu De Bordeaux - Hôpital Haut Lévêque, Pessac
- Germany (8):
  - Klinikum der Johann-Wolfgang Goethe, Universitaet Frankfurt am Main, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover, Lower Saxony
  - Friedrich-Alexander-Uniersitat Erlangen, Erlangen, QLD
  - CHARITÉ, Campus Virchow Klinikum, Berlin
  - Univeritatsklinikum Hamburg Eppendorf, Medizinische Klinik und Poliklinik, Hamburg
  - Universitaetsklinikum Heidelberg Medizinische Universitaetsklinik, Heidelberg
  - Universität Leipzig KöR, Medizinische Fakultät, Leipzig
  - University of Munich, LMU Klinikum Grosshadern, Munich
- Hong Kong (5):
  - Queen Mary Hospital, Hong Kong, Pokfulam
  - Prince Of Wales Hospital, Hong Kong, Shatin
  - Tuen Mun Hospital, Hong Kong, Tuen Mun, New Territories
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Humanity & Health Research Centre, Hong Kong
- Hungary (3):
  - Békés Megyei Kozponti Korhaz - Dr. Rethy Pal Tagkorhaz, Békéscsaba
  - Szent János Hospital, Budapest
  - University Of Debrecen, Department Of Medicine, Division Of Gastroenterology, Debrecen
- Israel (7):
  - Hadassah Hebrew University Medical Center, Jerusalem, Nazareth Elit
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Tel-Aviv Medical Center, Tel Aviv
- Italy (11):
  - Azienda Ospedaliero - Universitaria di Cagliari - Centro per lo Studio delle Malattie del Fegato, Monserrato, Cagliari
  - Università Politecnica delle Marche - Azienda Ospedaliero, Ancona
  - AOU Policlinico Sant' Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Sant´ Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Careggi Universita di Firenze, Florence
  - Azienda Socio-Sanitarla Territoriale (ASST) Santi Paolo e Carlo, Milan
  - AOU Ospedale Civile S. Agostino Estense - UO Medicina Metabolica, Modena
  - Azienda Socio Sanitaria Territoriale (ASST) di Monza, Monza
  - Azienda Ospedaliero - Universita di Padova, Padua
  - AOU Policlinico Paolo Giaccone - Di.Bi.M.I.S, Palermo
  - Policlinico Universitario Agostino Gemelli - Universita Cattolica del Sacro Cuore, Rome
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences, Kauno klinikos, Kaunas
  - Vilnius University Hospital Santaros klinikos, Vilnius
- Mexico (3):
  - Departamento De Gastroenterologia. Instituto Nacional De Ciencias Medicas Y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Medica Sur, S.A.B. de C.V., Mexico City, Mexico City
  - Consultorio Médico de la Dra Alma Laura Ladrón de Guevara Cetina, Mexico City, Mexico City
- Netherlands (5):
  - Radboud UMC, Nijmegen, Gelderland
  - Vrije Universiteit Medisch Centrum (VUMC), Amsterdam, North Holland
  - Erasmus Mc, Rotterdam, South Holland
  - Amsterdam University Medical Centre (AMC), Amsterdam
  - University Medical Center Utrecht, Utrecht
- New Zealand (2):
  - NZ Liver Transplant Unit, Auckland Hospital, Grafton, Auckland
  - Gastroenterology, Christchurch Hospital, Christchurch, Canterbury
- Poland (6):
  - Nzoz Vitamed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. J. Gromkowskiego, Pierwszy Oddzial Chorob Zakaznych, Wroclaw, Lover Silesia
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej - Curie, Klinika Gastroenterologii Onkologicznej, Warsaw, Masovian Voivodeship
  - Medical University of Warsaw Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie (SPCSK in Warsaw, Warsaw, Masovia
  - Oddział Gastr. I Hepat. Uniwersyteckie Centrum Kliniczne Im. Prof. K. Gibińskiego Sum, Katowice, Silesian Voivodeship
  - Dep. Of Gastroenterology UM Lublin, Lublin
- Centro Hospitalar Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon, Portugal
- Serbia (2):
  - Clinic For Gastroenterology And Hepatology Clinical Center Of Serbia, Belgrade
  - Clinical Hospital Centre Zvezdara, Belgrade
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan, Busanjin-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-Gu
  - Pusan National University Hospital, Busan, Seo-gu
- Spain (7):
  - Hospital Universitario Marqués De Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta De Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Virgen De La Victoria University Hospital, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - La Fe, Hospital ( Valence ), Valencia
- Sweden (2):
  - Karolinska University Hospital, Stockholm, Huddinge
  - Sahlgrenska Universitetssjukhuset, Gothenburg
- Switzerland (3):
  - Inselspital, University Of Bern, UVCM, DMLL, Bern
  - Kantonsspital St. Gallen, Clinic for Gastroeterologie and Hepatologie, Sankt Gallen
  - USZ, Klinik für Gastroenterologie und Hepatologie, Zurich
- Turkey (Türkiye) (2):
  - Ankara University School of Medicine Gastroenterology Dept., Ankara
  - Ege University School of Medicine Gastroenterology Dept., Izmir
- United Kingdom (9):
  - University Hospitals Bristol NHS Foundation Trust, Bristol, Avon
  - Plymouth Hospitals NHS Trust, Derriford Hospital, Plymouth, Devon
  - Gartnavel General Hospital, Glasgow, Lanarkshire
  - Forth Valley Royal Hospital, Larbert, Scotland
  - Institute of Cellular Medicine, Newcastle upon Tyne, Tyne and Wear
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Cambrigde University Hospitals NHS Foundation Trust, Cambridge
  - The Royal Free Hospital, London
  - Nottingham University Hospital Nhs Trust, Nottingham

REFERENCES:
- [Background] Lindor KD, Gershwin ME, Poupon R, Kaplan M, Bergasa NV, Heathcote EJ; American Association for Study of Liver Diseases. Primary biliary cirrhosis. Hepatology. 2009 Jul;50(1):291-308. doi: 10.1002/hep.22906. No abstract available. PMID 19554543
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. J Hepatol. 2009 Aug;51(2):237-67. doi: 10.1016/j.jhep.2009.04.009. Epub 2009 Jun 6. No abstract available. PMID 19501929
- [Derived] Kowdley KV, Hirschfield GM, Coombs C, Malecha ES, Bessonova L, Li J, Rathnayaka N, Mells G, Jones DE, Trivedi PJ, Hansen BE, Smith R, Wason J, Hiu S, Kareithi DN, Mason AL, Bowlus CL, Muller K, Carbone M, Berenguer M, Milkiewicz P, Adekunle F, Villamil A. COBALT: A Confirmatory Trial of Obeticholic Acid in Primary Biliary Cholangitis With Placebo and External Controls. Am J Gastroenterol. 2025 Feb 1;120(2):390-400. doi: 10.14309/ajg.0000000000003029. Epub 2024 Aug 14. PMID 39140490

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 334 participants were randomized into the study. The study was terminated early as the Data Monitoring Committee made the recommendation not to pursue further enrollment, given the lack of feasibility for this post-marketing study as designed. At termination, the study randomized <80% of planned enrollment.
Groups:
- Obeticholic Acid: Participants received obeticholic acid (OCA) 5 mg for a minimum of 3 months and titrating up to 10 mg for the remainder of the study (based on tolerability and Child-Pugh [CP] Score).
  Non-cirrhotic and classified as CP Class A: 5 mg tablet of OCA once daily, titrating up to a maximum of 10 mg OCA once daily based on tolerability at 3 months for the duration of the study (majority of participants).
  Cirrhotic and classified as CP Class B and C: 5 mg tablet of OCA once weekly for at least 3 months, titrating up to a maximum dose and frequency of 10 mg twice weekly based on tolerability and biochemical response for the duration of the study.
- Placebo: Participants received one tablet daily (or a lower frequency depending on CP score) for the remainder of the study.
Period: Overall Study
Arm/Group | Obeticholic Acid | Placebo
Started | 168 | 166
Received at Least 1 Dose of Study Drug | 168 | 166
Completed (The discontinuation reasons from here onward reflect discontinuation for withdrawal from study visits only. Reasons for discontinuation from study IP and reasons for discontinuation from study follow-up (phone call / medical record review) were also collected but are not reported here.) | 0 | 0
Not Completed | 168 | 166
Not completed — Adverse Event | 31 | 19
Not completed — Death | 9 | 6
Not completed — Lost to Follow-up | 2 | 7
Not completed — Physician Decision | 6 | 17
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 28 | 38
Not completed — Study Terminated by Sponsor | 72 | 61
Not completed — Initiated Commercial OCALIVA | 6 | 8
Not completed — Site Closure | 3 | 3
Not completed — Non-compliance with Study Drug | 3 | 1
Not completed — COVID-19 Pandemic Limitation | 2 | 0
Not completed — Liver Transplant | 3 | 3
Not completed — Liver Transplant Waitlist | 2 | 2
Not completed — Early Termination As Subject Was Randomized Without Meeting All Eligibility Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of the study drug.
Groups:
- Obeticholic Acid: Participants received OCA 5 mg for a minimum of 3 months and titrating up to 10 mg for the remainder of the study (based on tolerability and CP Score).
  Non-cirrhotic and classified as CP Class A: 5 mg tablet of OCA once daily, titrating up to a maximum of 10 mg OCA once daily based on tolerability at 3 months for the duration of the study (majority of participants).
  Cirrhotic and classified as CP Class B and C: 5 mg tablet of OCA once weekly for at least 3 months, titrating up to a maximum dose and frequency of 10 mg twice weekly based on tolerability and biochemical response for the duration of the study.
- Total: Total of all reporting groups
Arm/Group | Obeticholic Acid | Placebo | Total
Number analyzed (Participants) | 168 | 166 | 334
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 140 | 140 | 280
  >=65 years | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.28) | 53.9 (10.41) | 53.7 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 149 | 300
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 18 | 42
  Not Hispanic or Latino | 138 | 139 | 277
  Unknown or Not Reported | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 11 | 9 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 146 | 143 | 289
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Occurrence of Composite Endpoint
Description: To assess the effect of OCA, compared to placebo in conjunction with the established local standard of care, on clinical outcomes in participants with PBC as measured by time to the first occurrence of any of the following adjudicated events, derived as a composite event endpoint of death, liver transplant, model of end-stage liver disease (MELD) ≥15, uncontrolled ascites, or hospitalization for new onset or recurrence of variceal bleed, hepatic encephalopathy (as defined by a West Haven score of >=2), or spontaneous bacterial peritonitis. The clinical events distribution was estimated using the Kaplan-Meier methodology. Point estimates and 95% confidence intervals (CIs) for the clinical events distribution percentiles (25th and 50th) are provided.
Time Frame: Time to first occurrence from date of randomization until the time to accrue approximately 127 primary endpoint events (up to 7 years)
Population: The Intent-to-Treat (ITT) population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
days
  25th Percentile | 1092 [670 to 1464] | 970 [688 to 1342]
  50th Percentile | NA [1910 to NA] — NA= Not calculable due to insufficient clinical events. The upper 95% CI limit was not estimable due to an insufficient number of participants with clinical events, as indicated by NA. | NA [NA to NA] — NA= Not calculable due to insufficient clinical events. The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with clinical events, as indicated by NA.
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.954, Log Rank — Log rank p-value and hazard ratio are based on stratified analyses, with the randomization stratification factors entered in the interactive web response system (IWRS) as strata; Hazard Ratio, log = 1.01, 95% CI 2-sided [0.68 to 1.51]

2. Primary Outcome: Time to the First Occurrence of Primary Clinical Event (Expanded Endpoint)
Description: Primary clinical outcome event is the first occurrence of the following events: death, liver transplant, MELD score >=15 (MELD-Na score >=12 baseline), MELD-Na score >=15 (MELD-Na score <12 baseline), hospitalization for new onset or recurrence of variceal bleed, hepatic encephalopathy, spontaneous bacterial peritonitis (confirmed by diagnostic paracentesis), or bacterial empyema, uncontrolled or refractory ascites (requiring large volume paracentesis), portal hypertension syndromes, progression to decompensated liver disease, and progression to clinical evidence of portal hypertension without decompensation (for participants without decompensation or clinical evidence of portal hypertension at baseline). 71 endpoint events were observed in the OCA arm, and 80 were observed in the Placebo arm. The clinical events distribution was estimated using the Kaplan-Meier methodology. Point estimates and 95% CIs for the clinical events distribution percentiles (25th and 50th) are provided.
Time Frame: as for outcome 1
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
days
  25th Percentile | 370 [261 to 638] | 450 [358 to 569]
  50th Percentile | 1827 [1198 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with clinical events, as indicated by NA | 1102 [841 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with clinical events, as indicated by NA
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.304, Log Rank — Log rank p-value and hazard ratio are based on stratified analyses, with the randomization stratification factors entered in the IWRS as strata; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.61 to 1.16]

3. Secondary Outcome: Time To First Occurrence Of Severe Decompensating Events of Expanded Composite Endpoint
Description: The first occurrence of the key secondary clinical event refers to the first occurrence of the following events: death, liver transplant, MELD-Na score >=15 if MELD-Na< 12 at baseline, MELD score >=15 if MELD-Na >=12 at baseline, uncontrolled or refractory ascites, portal hypertension syndromes (hepatorenal syndrome, portopulmonary syndrome, hepatopulmonary syndrome) or hospitalization for new onset or recurrence of variceal bleed, hepatic encephalopathy, spontaneous bacterial peritonitis, or bacterial empyema. The clinical events distribution was estimated using the Kaplan-Meier methodology. Point estimates and 95% CIs for the clinical events distribution percentiles (25th and 50th) are provided.
Time Frame: Time to first occurrence from date of randomization until the date of first documented progression or date of death from any cause, whichever came first (up to 7 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
days
  25th Percentile | 1092 [670 to 1408] | 929 [679 to 1342]
  50th Percentile | NA [1910 to NA] — NA= Not calculable due to insufficient clinical events. The upper 95% CI limit was not estimable due to an insufficient number of participants with clinical events, as indicated by NA. | NA [NA to NA] — NA= Not calculable due to insufficient clinical events. The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with clinical events, as indicated by NA.
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.898, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.69 to 1.52]

4. Secondary Outcome: Time To Liver Transplant Or Death (All-cause)
Description: The effect of OCA compared to placebo on time to liver transplant or death (all-cause) was assessed. The events distribution was estimated using the Kaplan-Meier methodology. Point estimates and 95% CIs for the clinical events distribution percentiles (25th and 50th) are provided.
Time Frame: Time to first occurrence from date of randomization until the date of first documented liver transplant or date of death from any cause (up to 7 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
days
  25th Percentile | 1580 [1275 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA. | 1803 [1206 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA.
  50th Percentile | NA [NA to NA] — NA= Not calculable due to insufficient events The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with events, as indicated by NA. | NA [NA to NA] — NA= Not calculable due to insufficient events The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with events, as indicated by NA.
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.594, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.69 to 1.91]

5. Secondary Outcome: Time to First Occurrence of Fatal Event (All-Cause)
Description: The results represent the ratio of OCA to placebo. The fatal events distribution was estimated using the Kaplan-Meier methodology. Point estimates and 95% CIs for the fatal events distribution percentiles (25th and 50th) are provided
Time Frame: Time to first occurrence from date of randomization until the date of death from any cause (up to 7 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
days
  25th Percentile | NA [NA to NA] — NA= Not calculable due to insufficient fatal events. The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with fatal events, as indicated by NA. | NA [NA to NA] — NA= Not calculable due to insufficient fatal events. The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with fatal events, as indicated by NA.
  50th Percentile | NA [NA to NA] — NA= Not calculable due to insufficient fatal events. The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with fatal events, as indicated by NA. | NA [NA to NA] — NA= Not calculable due to insufficient fatal events. The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with fatal events, as indicated by NA.
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.568, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.57 to 2.78]

6. Secondary Outcome: Time to First Occurrence of Liver Transplant
Description: The effect of OCA compared to placebo on time to occurrence of a liver transplant was assessed. The results represented the ratio of OCA to placebo. A hazard ratio <1 indicated an advantage for OCA. The event of interest was summarized through Cumulative Incidence Function (CIF) estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of first documented liver transplant or date of death from any cause (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0.18 [0.11 to 0.26] | 0.16 [0.09 to 0.23]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.769, Gray's Test — Gray's test p-value and hazard ratio are based on stratified analyses, with the randomization stratification factors entered in the interactive web response system (IWRS) as strata; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.59 to 2.07]

7. Secondary Outcome: Time to First Occurrence of Hospitalization Due to Hepatic Events
Description: Hospitalization events include new onset or recurrent variceal bleed, hepatic encephalopathy (as defined by a West Haven score of >=2), spontaneous bacterial peritonitis (confirmed by diagnostic paracentesis OR presence of >250/mm^3 polymorph leucocytes [PMNs] in the ascitic fluid), bacterial empyema is confirmed by diagnostic thoracentesis OR presence of >250/mm^3 PMNs in the pleural fluid. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of hospitalization, liver transplant or death from any cause, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0.11 [0.06 to 0.17] | 0.18 [0.10 to 0.26]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.599, Gray's Test — Gray's test p-value and hazard ratio are based on stratified analyses, with the randomization stratification factors entered in the IWRS as strata; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.42 to 1.67]

8. Secondary Outcome: Time to First Occurrence of Uncontrolled or Refractory Ascites
Description: Uncontrolled or refractory ascites are defined as diuretic-resistant ascites requiring large-volume paracentesis. The effect of OCA compared to placebo on time to the first occurrence of uncontrolled or refractory ascites was assessed. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of first documented uncontrolled or refractory ascites, liver transplant or date of death from any cause, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0.02 [0.01 to 0.05] | 0.04 [0.01 to 0.08]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.745, Gray's Test — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.18 to 3.43]

9. Secondary Outcome: Time to First Occurrence of MELD Score ≥15
Description: The MELD score is useful in assessing participants with significant decompensation. The MELD score is now used by the United Network for Organ Sharing in the United States and Eurotransplants to manage organ allocation for liver transplantation. The MELD score is derived from the participant's serum total bilirubin, serum creatinine, and International Normalized Ratio (INR), as appropriate, to predict survival. The MELD score ranges from 6 to 40. The higher the score, the more likely a participant will receive a liver from a deceased donor when an organ becomes available. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of first documented MELD Score ≥15, liver transplant or date of death from any cause, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0.13 [0.07 to 0.19] | 0.18 [0.11 to 0.25]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.437, Gray's Test — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.43 to 1.44]

10. Secondary Outcome: Time To Development Of Varix/Varices
Description: The effect of OCA compared to placebo on time to development of varix/varices was assessed. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of first documented development of varix/varices, liver transplant or death from any cause, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0.07 [0.03 to 0.12] | 0.09 [0.04 to 0.17]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.838, Gray's Test — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.37 to 2.24]

11. Secondary Outcome: Time To Liver-Related Death
Description: The effect of OCA compared to placebo on time to liver-related death was assessed. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of first liver-related or non-liver- related death, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0.03 [0.01 to 0.07] | 0.04 [0.01 to 0.09]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.980, Gray's Test — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.26 to 4.04]

12. Secondary Outcome: Time To Liver-Related Death Or Liver Transplant
Description: The effect of OCA compared to placebo on time to liver-related death or liver transplant was assessed. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of liver transplant, liver-related death or non-liver-related death from any cause, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0.20 [0.13 to 0.29] | 0.19 [0.12 to 0.27]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.933, Gray's Test — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.58 to 1.83]

13. Secondary Outcome: Time To Liver-Related Death, Liver Transplant, Or MELD Score ≥15
Description: The effect of OCA compared to placebo on time to liver-related death, liver transplant, or MELD Score ≥15 was assessed. The MELD score is useful in assessing participants with significant decompensation. The MELD score is now used by the United Network for Organ Sharing in the United States and Eurotransplants to manage organ allocation for liver transplantation. The MELD score is derived from the participant's serum total bilirubin, serum creatinine, and INR, as appropriate, to predict survival. The MELD score ranges from 6 to 40. The higher the score, the more likely a participant will receive a liver from a deceased donor when an organ becomes available. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of liver transplant, liver-related death, non-liver-related death from any cause or MELD Score ≥15, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0.25 [0.17 to 0.33] | 0.29 [0.21 to 0.37]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.468, Gray's Test — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.53 to 1.34]

14. Secondary Outcome: Progression To Cirrhosis (for Noncirrhotic Subjects at Baseline)
Description: When a participant is identified as noncirrhotic at the Baseline and exhibited any signs or symptoms associated with progression to cirrhosis, the participant was assessed by Fibroscan® TE where available. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of cirrhosis, liver transplant or death from any cause, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 78 | 62
proportion of participants | 0.07 [0.02 to 0.16] | 0.15 [0.06 to 0.27]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.178, Gray's Test — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.13 to 1.41]
Statistical Analysis 2: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.190, Cochran-Mantel-Haenszel; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.13 to 1.41]

15. Secondary Outcome: Time To Occurrence Of Hepatocellular Carcinoma (HCC)
Description: The effect of OCA compared to placebo on time to occurrence of HCC was assessed. The event of interest was summarized through CIF estimate at 5 years.
Time Frame: Time to first occurrence from date of randomization until the date of HCC diagnosis, liver transplant or death from any cause, whichever came first (up to 5 years)
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
proportion of participants | 0 [NA to NA] — The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with events, as indicated by NA. | 0.01 [0 to 0.05]
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority; p = 0.443, Gray's Test — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.05 to 3.54]

16. Secondary Outcome: Change From Baseline To Month 24 Of Total Bilirubin
Description: Liver biochemistry, which includes total bilirubin, was assessed to evaluate biochemical triggers that would prompt an immediate reevaluation of participants for potential hepatic injury or hepatic decompensation. Analysis was performed using mixed model repeated measures (MMRM), including treatment group, time, treatment group by time interaction, and randomization stratification factors as entered in the IWRS as fixed effects and baseline values as a covariate.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
mg/dL
  Month 6: number analyzed (Participants) | 149 | 153
  Month 6 | 0.10 (0.069) | 0.17 (0.069)
  Month 12: number analyzed (Participants) | 126 | 138
  Month 12 | 0.26 (0.113) | 0.29 (0.111)
  Month 24: number analyzed (Participants) | 97 | 101
  Month 24 | 0.30 (0.141) | 0.63 (0.138)

17. Secondary Outcome: Change From Baseline To Month 24 Of Direct Bilirubin
Description: Liver biochemistry, which includes direct bilirubin, was assessed to evaluate biochemical triggers that would prompt an immediate reevaluation of participants for potential hepatic injury or hepatic decompensation. Analysis was performed using MMRM, including treatment group, time, treatment group by time interaction, and randomization stratification factors as entered in the IWRS as fixed effects and baseline values as a covariate.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
mg/dL
  Month 6: number analyzed (Participants) | 147 | 147
  Month 6 | 0.11 (0.054) | 0.14 (0.054)
  Month 12: number analyzed (Participants) | 121 | 138
  Month 12 | 0.13 (0.073) | 0.22 (0.071)
  Month 24: number analyzed (Participants) | 96 | 97
  Month 24 | 0.19 (0.107) | 0.48 (0.106)

18. Secondary Outcome: Change From Baseline To Month 24 Of Aspartate Aminotransferase (AST)
Description: Liver biochemistry, which includes AST, was assessed to evaluate biochemical triggers that would prompt an immediate reevaluation of participants for potential hepatic injury or hepatic decompensation. Analysis was performed using MMRM, including treatment group, time, treatment group by time interaction, and randomization stratification factors as entered in the IWRS as fixed effects and baseline values as a covariate.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
U/L
  Month 6: number analyzed (Participants) | 147 | 150
  Month 6 | -14.5 (2.21) | -0.6 (2.19)
  Month 12: number analyzed (Participants) | 124 | 138
  Month 12 | -11.8 (2.36) | -5.4 (2.27)
  Month 24: number analyzed (Participants) | 97 | 102
  Month 24 | -14.8 (2.78) | -6.0 (2.72)

19. Secondary Outcome: Change From Baseline To Month 24 Of Alanine Aminotransferase (ALT)
Description: Liver biochemistry, which includes ALT, was assessed to evaluate biochemical triggers that would prompt an immediate reevaluation of participants for potential hepatic injury or hepatic decompensation. Analysis was performed using MMRM, including treatment group, time, treatment group by time interaction, and randomization stratification factors as entered in the IWRS as fixed effects and baseline values as a covariate.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
U/L
  Month 6: number analyzed (Participants) | 149 | 153
  Month 6 | -24.3 (2.62) | -7.4 (2.59)
  Month 12: number analyzed (Participants) | 126 | 138
  Month 12 | -20.5 (3.49) | -12.8 (3.37)
  Month 24: number analyzed (Participants) | 97 | 100
  Month 24 | -28.5 (2.92) | -19.4 (2.87)

20. Secondary Outcome: Change From Baseline To Month 24 Of Alkaline Phosphatase (ALP)
Description: Liver biochemistry, which includes ALP, was assessed to evaluate biochemical triggers that would prompt an immediate reevaluation of participants for potential hepatic injury or hepatic decompensation. Analysis was performed using MMRM, including treatment group, time, treatment group by time interaction, and randomization stratification factors as entered in the IWRS as fixed effects and baseline values as a covariate.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
U/L
  Month 6: number analyzed (Participants) | 150 | 152
  Month 6 | -134.3 (10.86) | -37.4 (10.85)
  Month 12: number analyzed (Participants) | 126 | 138
  Month 12 | -144.8 (12.05) | -68.8 (11.72)
  Month 24: number analyzed (Participants) | 98 | 102
  Month 24 | -156.4 (14.93) | -113.1 (14.60)

21. Secondary Outcome: Change From Baseline To Month 24 Of Gamma-glutamyl Transferase (GGT)
Description: Liver biochemistry, which includes GGT, was assessed to evaluate biochemical triggers that would prompt an immediate reevaluation of participants for potential hepatic injury or hepatic decompensation. Analysis was performed using MMRM, including treatment group, time, treatment group by time interaction, and randomization stratification factors as entered in the IWRS as fixed effects and baseline values as a covariate.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
U/L
  Month 6: number analyzed (Participants) | 150 | 152
  Month 6 | -155.5 (15.04) | -47.0 (14.99)
  Month 12: number analyzed (Participants) | 126 | 138
  Month 12 | -152.2 (18.24) | -63.4 (17.71)
  Month 24: number analyzed (Participants) | 98 | 102
  Month 24 | -175.6 (22.49) | -127.7 (22.04)

22. Secondary Outcome: Change From Baseline To Month 24 Of Albumin
Description: Liver biochemistry, which includes albumin, was assessed to evaluate biochemical triggers that would prompt an immediate reevaluation of participants for potential hepatic injury or hepatic decompensation. Analysis was performed using MMRM, including treatment group, time, treatment group by time interaction, and randomization stratification factors as entered in the IWRS as fixed effects and baseline values as a covariate.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
g/L
  Month 6: number analyzed (Participants) | 150 | 153
  Month 6 | -0.4 (0.19) | -0.1 (0.19)
  Month 12: number analyzed (Participants) | 126 | 138
  Month 12 | -0.3 (0.23) | -0.3 (0.22)
  Month 24: number analyzed (Participants) | 98 | 102
  Month 24 | -0.1 (0.29) | -1.1 (0.28)

23. Secondary Outcome: Change From Baseline To Month 24 Of INR
Description: The coagulation test, which includes INR, was assessed to evaluate biochemical triggers that would prompt an immediate reevaluation of participants for potential hepatic injury or hepatic decompensation. INR is the ratio of tested prothrombin time to normal prothrombin time, to a power designated the international sensitivity index (ISI). INR normal range is 0.8 to 1.2 (female and male). Analysis was performed using MMRM, including treatment group, time, treatment group by time interaction, and randomization stratification factors as entered in the IWRS as fixed effects and baseline values as a covariate.
Time Frame: Baseline up to Month 24
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
ratio
  Month 6: number analyzed (Participants) | 148 | 146
  Month 6 | 0.02 (0.014) | 0.02 (0.014)
  Month 12: number analyzed (Participants) | 124 | 136
  Month 12 | 0.01 (0.009) | 0.02 (0.008)
  Month 24: number analyzed (Participants) | 93 | 98
  Month 24 | 0.03 (0.014) | 0.06 (0.014)

24. Secondary Outcome: Change From Baseline To Month 72 Of MELD Score
Description: The MELD score is useful in assessing participants with significant decompensation. The MELD score is now used by the United Network for Organ Sharing in the United States and Eurotransplants to manage organ allocation for liver transplantation. The MELD score is derived from the participant's serum total bilirubin, serum creatinine, and INR, as appropriate, to predict survival. The MELD score ranges from 6 to 40. The higher the score, the more likely a participant will receive a liver from a deceased donor when an organ becomes available.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
score on a scale
  Month 12: number analyzed (Participants) | 121 | 134
  Month 12 | 0 [-0.60 to 0.60] | 0 [-0.50 to 1.30]
  Month 24: number analyzed (Participants) | 91 | 97
  Month 24 | 0 [-1.00 to 0.70] | 0.20 [-0.50 to 1.70]
  Month 36: number analyzed (Participants) | 71 | 59
  Month 36 | 0 [-1.00 to 0.50] | 0.60 [-0.50 to 2.90]
  Month 48: number analyzed (Participants) | 48 | 34
  Month 48 | 0 [-0.95 to 1.45] | 0.40 [-0.80 to 1.60]
  Month 60: number analyzed (Participants) | 31 | 20
  Month 60 | 0 [-1.30 to 0.40] | 0 [-1.20 to 1.85]
  Month 72: number analyzed (Participants) | 7 | 4
  Month 72 | 0 [-1.20 to 5.20] | 1.95 [-1.40 to 3.10]

25. Secondary Outcome: Change From Baseline To Month 72 Of MELD-Na Score
Description: The MELD-Na score is another useful predictor in assessing participants with significant decompensation. The MELD-Na took into account the effect of serum sodium as a reflection of renal function and hypothetically may improve the accuracy of the model score. The MELD-Na score is derived from the participant's serum total bilirubin, serum creatinine, INR, and serum sodium, as appropriate, to predict survival. The MELD-Na score ranges from 6 to 40. The higher the score, the more likely a participant will receive a liver from a deceased donor when an organ becomes available.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
score on a scale
  Month 12: number analyzed (Participants) | 121 | 132
  Month 12 | 0 [-1.0 to 1.0] | 0 [-1.0 to 1.0]
  Month 24: number analyzed (Participants) | 91 | 97
  Month 24 | 0 [-2.0 to 0] | 0 [-1.0 to 1.0]
  Month 36: number analyzed (Participants) | 71 | 59
  Month 36 | 0 [-2.0 to 0] | 0 [-1.0 to 2.0]
  Month 48: number analyzed (Participants) | 48 | 34
  Month 48 | 0 [-2.0 to 2.0] | 0 [-2.0 to 2.0]
  Month 60: number analyzed (Participants) | 31 | 20
  Month 60 | -1.0 [-3.0 to 0] | 0 [-2.5 to 1.5]
  Month 72: number analyzed (Participants) | 6 | 4
  Month 72 | 0 [-2.0 to 0] | 0.5 [-3.5 to 1.5]

26. Secondary Outcome: Change From Baseline To Month 72 Of CPS
Description: Child-Pugh Score (Pugh 1973, Lucey 1997) was calculated and reported within the electronic data capture (EDC) system based on data entered into the CRF by adding the scores from the 5 factors and could have ranged from 5 to15. A total score of 5 to 6 was considered Grade A (mild, well-compensated disease); 7 to 9 was Grade B (moderate, significant functional compromise); and 10 and above was Grade C (severe, decompensated disease).
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
score on a scale
  Month 12: number analyzed (Participants) | 126 | 135
  Month 12 | 0 [0 to 0] | 0 [0 to 1.0]
  Month 24: number analyzed (Participants) | 93 | 97
  Month 24 | 0 [0 to 0] | 0 [0 to 1.0]
  Month 36: number analyzed (Participants) | 71 | 57
  Month 36 | 0 [0 to 0] | 0 [0 to 1.0]
  Month 48: number analyzed (Participants) | 47 | 35
  Month 48 | 0 [0 to 0] | 0 [0 to 1.0]
  Month 60: number analyzed (Participants) | 31 | 20
  Month 60 | 0 [0 to 0] | 0 [0 to 1.0]
  Month 72: number analyzed (Participants) | 7 | 4
  Month 72 | 0 [0 to 2.0] | 1.0 [0 to 1.0]

27. Secondary Outcome: Change From Baseline To Month 72 Of Mayo Risk Score (MRS)
Description: Mayo Risk Score (MRS) was calculated and reported within the EDC system. Calculation of MRS included Investigator assessment of peripheral edema and the use of diuretic therapy, which was assessed during the adverse event and concomitant medicine review at the scheduled visits and entered into the CRF, as well as total bilirubin, albumin, and prothrombin time results obtained from the central laboratory data. There is no maximum and minimum range of score but an increase in the MRS represents an increase in the risk of death.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
score on a scale
  Month 12: number analyzed (Participants) | 117 | 128
  Month 12 | 0 [-0.380 to 0.320] | 0.080 [-0.205 to 0.535]
  Month 24: number analyzed (Participants) | 80 | 91
  Month 24 | -0.080 [-0.270 to 0.390] | 0.140 [-0.170 to 0.660]
  Month 36: number analyzed (Participants) | 65 | 53
  Month 36 | -0.040 [-0.410 to 0.280] | 0.050 [-0.240 to 0.650]
  Month 48: number analyzed (Participants) | 43 | 29
  Month 48 | 0.030 [-0.430 to 0.620] | 0.210 [-0.240 to 0.810]
  Month 60: number analyzed (Participants) | 28 | 18
  Month 60 | -0.145 [-0.575 to 0.160] | -0.060 [-0.490 to 0.790]
  Month 72: number analyzed (Participants) | 6 | 4
  Month 72 | -0.130 [-0.460 to 0.320] | 0.990 [0.240 to 1.165]

28. Secondary Outcome: Change From Baseline To Month 72 Of Immunoglobulin-M (IgM)
Description: Markers of inflammation, which include IgM, were assessed.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
g/L
  Month 12: number analyzed (Participants) | 124 | 135
  Month 12 | -0.305 [-0.955 to 0.025] | -0.160 [-0.720 to 0.200]
  Month 24: number analyzed (Participants) | 97 | 101
  Month 24 | -0.470 [-1.250 to -0.090] | -0.230 [-0.630 to 0.170]
  Month 36: number analyzed (Participants) | 72 | 59
  Month 36 | -0.700 [-1.440 to -0.025] | -0.330 [-1.270 to 0]
  Month 48: number analyzed (Participants) | 48 | 35
  Month 48 | -0.525 [-1.615 to 0.005] | -0.690 [-1.540 to 0.090]
  Month 60: number analyzed (Participants) | 32 | 21
  Month 60 | -0.745 [-1.545 to -0.075] | -0.350 [-1.050 to -0.150]
  Month 72: number analyzed (Participants) | 7 | 4
  Month 72 | -1.590 [-4.100 to 0.050] | -0.640 [-1.060 to 0.645]

29. Secondary Outcome: Change From Baseline To Month 72 Of C-reactive Protein (CRP)
Description: Markers of inflammation, which include CRP, were assessed.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
mg/L
  Month 12: number analyzed (Participants) | 127 | 137
  Month 12 | -0.140 [-1.320 to 1.360] | 0.400 [-0.760 to 2.720]
  Month 24: number analyzed (Participants) | 98 | 101
  Month 24 | -0.280 [-1.210 to 1.110] | 0.290 [-1.450 to 2.950]
  Month 36: number analyzed (Participants) | 74 | 59
  Month 36 | -0.525 [-2.160 to 0.630] | 0.340 [-1.460 to 3.830]
  Month 48: number analyzed (Participants) | 51 | 36
  Month 48 | -0.260 [-1.700 to 2.180] | -0.180 [-1.200 to 2.025]
  Month 60: number analyzed (Participants) | 33 | 22
  Month 60 | -0.720 [-3.020 to 0.740] | -0.730 [-2.700 to 1.650]
  Month 72: number analyzed (Participants) | 7 | 4
  Month 72 | -0.100 [-2.740 to 2.570] | 0.765 [-2.630 to 4.715]

30. Secondary Outcome: Change From Baseline To Month 72 Of Tumor Necrosis Factor-α (TNF-α)
Description: Markers of inflammation, which include TNF-α, were assessed.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
pg/mL
  Month 12: number analyzed (Participants) | 117 | 123
  Month 12 | 0 [-0.362 to 0.580] | 0.058 [-0.236 to 0.791]
  Month 24: number analyzed (Participants) | 91 | 95
  Month 24 | 0.203 [-0.213 to 0.758] | 0.323 [-0.039 to 0.654]
  Month 36: number analyzed (Participants) | 66 | 56
  Month 36 | 0.055 [-0.304 to 0.627] | 0.296 [-0.078 to 0.750]
  Month 48: number analyzed (Participants) | 46 | 33
  Month 48 | 0.165 [-0.195 to 0.814] | 0.539 [0.113 to 0.918]
  Month 60: number analyzed (Participants) | 29 | 19
  Month 60 | -0.009 [-0.765 to 0.596] | 0.419 [-0.153 to 0.753]
  Month 72: number analyzed (Participants) | 6 | 3
  Month 72 | 0.046 [-0.390 to 0.175] | 0.616 [-1.318 to 0.788]

31. Secondary Outcome: Change From Baseline To Month 72 Of Fibroblast Growth Factor-19 (FGF-19)
Description: Markers of hepatic fibrosis, which include FGF-19, were assessed.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
pg/mL
  Month 12: number analyzed (Participants) | 124 | 132
  Month 12 | 73.50 [2.85 to 208.00] | -2.80 [-57.65 to 36.50]
  Month 24: number analyzed (Participants) | 95 | 97
  Month 24 | 72.00 [1.00 to 211.00] | -0.40 [-63.00 to 61.40]
  Month 36: number analyzed (Participants) | 69 | 59
  Month 36 | 39.90 [-17.70 to 132.00] | -2.00 [-51.00 to 50.80]
  Month 48: number analyzed (Participants) | 47 | 34
  Month 48 | 56.00 [-24.00 to 219.00] | -9.45 [-59.90 to 39.30]
  Month 60: number analyzed (Participants) | 31 | 22
  Month 60 | 14.40 [-30.00 to 183.00] | -1.45 [-83.40 to 156.00]
  Month 72: number analyzed (Participants) | 5 | 4
  Month 72 | -106.90 [-172.30 to -1.00] | -62.00 [-239.00 to -26.50]

32. Secondary Outcome: Change From Baseline To Month 72 Of Cytokeratin-18 (CK-18)
Description: Markers of inflammation, which include CK-18, were assessed.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
U/L
  Month 12: number analyzed (Participants) | 126 | 133
  Month 12 | -34.450 [-138.010 to 45.800] | 9.100 [-78.540 to 123.770]
  Month 24: number analyzed (Participants) | 97 | 100
  Month 24 | -57.660 [-158.960 to 8.470] | 17.545 [-54.630 to 165.835]
  Month 36: number analyzed (Participants) | 72 | 59
  Month 36 | -45.935 [-171.225 to 18.715] | 6.680 [-112.010 to 76.110]
  Month 48: number analyzed (Participants) | 50 | 35
  Month 48 | -81.035 [-158.900 to 33.550] | 0.290 [-130.710 to 79.410]
  Month 60: number analyzed (Participants) | 33 | 21
  Month 60 | -117.660 [-232.770 to 0] | -56.390 [-159.780 to 77.020]
  Month 72: number analyzed (Participants) | 7 | 4
  Month 72 | -182.590 [-207.020 to 17.060] | -32.745 [-199.555 to 78.070]

33. Secondary Outcome: Change From Baseline To Month 72 Of 7α-hydroxy-4-cholesten-3-one (C4)
Description: Markers of hepatic fibrosis, which include C4, were assessed.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
ng/mL
  Month 12: number analyzed (Participants) | 116 | 132
  Month 12 | -2.222 [-8.110 to 0.002] | -0.250 [-2.691 to 1.523]
  Month 24: number analyzed (Participants) | 96 | 98
  Month 24 | -3.700 [-10.119 to -0.885] | -0.861 [-5.500 to 0.900]
  Month 36: number analyzed (Participants) | 71 | 60
  Month 36 | -3.826 [-9.380 to 0.182] | -1.225 [-5.620 to 1.161]
  Month 48: number analyzed (Participants) | 49 | 34
  Month 48 | -4.220 [-9.870 to 0] | -1.168 [-12.240 to 1.691]
  Month 60: number analyzed (Participants) | 33 | 22
  Month 60 | -3.250 [-10.334 to -0.110] | -1.161 [-9.591 to 0.660]
  Month 72: number analyzed (Participants) | 7 | 4
  Month 72 | -7.500 [-10.914 to -0.690] | -0.947 [-15.281 to -0.277]

34. Secondary Outcome: Change From Baseline To Month 72 Of Enhanced Liver Fibrosis (ELF)
Description: Liver fibrosis was assessed using ELF test. The ELF test assessed: hyaluronic acid, procollagen3 N-terminal peptide, and a tissue inhibitor of metalloproteinase 1. The ELF test is a composite score: < 7.7: no to mild fibrosis; ≥ 7.7 - < 9.8: Moderate fibrosis; ≥ 9.8 - < 11.3: Severe fibrosis; ≥ 11.3: Cirrhosis. A negative change from Baseline suggests decreased fibrosis.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
score on a scale
  Month 12: number analyzed (Participants) | 126 | 127
  Month 12 | 0.10 [-0.50 to 0.60] | 0.10 [-0.20 to 0.70]
  Month 24: number analyzed (Participants) | 95 | 95
  Month 24 | 0 [-0.70 to 0.60] | 0.20 [-0.40 to 1.00]
  Month 36: number analyzed (Participants) | 71 | 59
  Month 36 | -0.20 [-0.90 to 0.70] | 0 [-0.60 to 0.70]
  Month 48: number analyzed (Participants) | 48 | 34
  Month 48 | 0.25 [-0.45 to 0.80] | 0.10 [-0.70 to 1.10]
  Month 60: number analyzed (Participants) | 33 | 21
  Month 60 | -0.20 [-1.20 to 0.60] | 0.10 [-1.00 to 1.00]
  Month 72: number analyzed (Participants) | 7 | 4
  Month 72 | 0 [-0.80 to 2.80] | -0.20 [-1.10 to 0.45]

35. Secondary Outcome: Change From Baseline To Month 72 Of Liver Stiffness - Transient Elastography
Description: Hepatic stiffness was measured using non-invasive transient Elastography with Fibroscan® TE device.
Time Frame: Baseline up to Month 72
Population: The ITT population included all randomized participants who received any dosage of OCA or placebo.
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
kPa
  Month 12: number analyzed (Participants) | 88 | 90
  Month 12 | 0.25 [-2.40 to 4.05] | 0.90 [-1.80 to 7.30]
  Month 24: number analyzed (Participants) | 67 | 67
  Month 24 | -0.60 [-2.60 to 3.60] | 1.50 [-2.20 to 15.60]
  Month 36: number analyzed (Participants) | 49 | 41
  Month 36 | 0.30 [-3.40 to 5.50] | 2.00 [-1.60 to 9.10]
  Month 48: number analyzed (Participants) | 31 | 19
  Month 48 | 0.70 [-2.20 to 4.00] | 1.00 [-2.80 to 11.90]
  Month 60: number analyzed (Participants) | 19 | 14
  Month 60 | 0.20 [-2.50 to 6.00] | -1.35 [-4.70 to 1.90]
  Month 72: number analyzed (Participants) | 5 | 3
  Month 72 | -2.40 [-2.50 to 2.70] | 3.20 [-2.20 to 8.70]

36. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (for example, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or procedure, whether or not considered related to the medicinal product or procedure, which occurred during the course of the clinical study. TEAEs were defined as AEs that occurred on or after the date and time of study drug administration, or those that first occurred before dosing but worsened in frequency or severity after study drug administration. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to the last IP dose plus 30 days and prior to commercial OCA initiation date (up to 7 years)
Population: The safety population consisted of all participants who received any amount of OCA or placebo. Treatment assignment based on the treatment received before any initiation of commercial OCA.
Measure: Number; unit: participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 168 | 166
participants
  TEAEs | 162 | 158
  SAEs | 53 | 53

37. Secondary Outcome: Pharmacokinetic (PK) Population: Fasting Trough Concentrations Of OCA By Dose Regimen
Description: The fasting trough PK concentrations of OCA of different dose regimens taken throughout the study are reported.
Time Frame: Months 3, 6, 9, 12, 24, 36, 48, and 60
Population: The PK Population included all OCA participants who had at least 1 confirmed fasted analyzable sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Obeticholic Acid: Participants who had at least 1 confirmed fasted analyzable OCA sample. Participants fasted for approximately 8 hours prior to the visit and had no major protocol deviations that potentially affected exposure levels.
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 149
ng/mL
  5 mg QD (Month 3): number analyzed (Participants) | 118
  5 mg QD (Month 3) | 119 (185)
  5 mg QD (Month 6): number analyzed (Participants) | 46
  5 mg QD (Month 6) | 102 (186)
  5 mg QD (Month 9): number analyzed (Participants) | 3
  5 mg QD (Month 9) | 175 (33.0)
  5 mg QD (Month 12): number analyzed (Participants) | 32
  5 mg QD (Month 12) | 117 (153)
  5 mg QD (Month 24): number analyzed (Participants) | 16
  5 mg QD (Month 24) | 113 (121)
  5 mg QD (Month 36): number analyzed (Participants) | 11
  5 mg QD (Month 36) | 84.5 (169)
  5 mg QD (Month 48): number analyzed (Participants) | 6
  5 mg QD (Month 48) | 203 (181)
  5 mg QD (Month 60): number analyzed (Participants) | 2
  5 mg QD (Month 60) | 7.96 (173)
  5 mg QOD (Month 3): number analyzed (Participants) | 9
  5 mg QOD (Month 3) | 123 (191)
  5 mg QOD (Month 6): number analyzed (Participants) | 8
  5 mg QOD (Month 6) | 103 (232)
  5 mg QOD (Month 9): number analyzed (Participants) | 1
  5 mg QOD (Month 9) | 396 (NA) — No variation was calculated.
  5 mg QOD (Month 12): number analyzed (Participants) | 7
  5 mg QOD (Month 12) | 103 (97.2)
  5 mg QOD (Month 24): number analyzed (Participants) | 3
  5 mg QOD (Month 24) | 134 (17.1)
  5 mg QOD (Month 48): number analyzed (Participants) | 1
  5 mg QOD (Month 48) | 307 (NA) — No variation was calculated.
  5 mg QW (Month 3): number analyzed (Participants) | 7
  5 mg QW (Month 3) | 57.3 (199)
  5 mg QW (Month 6): number analyzed (Participants) | 5
  5 mg QW (Month 6) | 31.0 (125)
  5 mg QW (Month 12): number analyzed (Participants) | 6
  5 mg QW (Month 12) | 73.5 (302)
  5 mg QW (Month 24): number analyzed (Participants) | 4
  5 mg QW (Month 24) | 171 (109)
  5 mg QW (Month 36): number analyzed (Participants) | 2
  5 mg QW (Month 36) | 245 (34.8)
  5 mg QW (Month 48): number analyzed (Participants) | 2
  5 mg QW (Month 48) | 141 (216)
  5 mg Q2W (Month 3): number analyzed (Participants) | 3
  5 mg Q2W (Month 3) | 61.9 (54.7)
  5 mg Q2W (Month 6): number analyzed (Participants) | 4
  5 mg Q2W (Month 6) | 108 (57.1)
  5 mg Q2W (Month 12): number analyzed (Participants) | 4
  5 mg Q2W (Month 12) | 187 (30.8)
  5 mg Q2W (Month 24): number analyzed (Participants) | 5
  5 mg Q2W (Month 24) | 208 (61.0)
  5 mg Q2W (Month 36): number analyzed (Participants) | 9
  5 mg Q2W (Month 36) | 225 (159)
  5 mg Q2W (Month 48): number analyzed (Participants) | 4
  5 mg Q2W (Month 48) | 502 (59.6)
  5 mg Q2W (Month 60): number analyzed (Participants) | 1
  5 mg Q2W (Month 60) | 7.32 (NA) — No variation was calculated.
  5 mg other regimens (Month 3): number analyzed (Participants) | 2
  5 mg other regimens (Month 3) | 50.3 (1730)
  5 mg other regimens (Month 6): number analyzed (Participants) | 2
  5 mg other regimens (Month 6) | 79.6 (68.2)
  5 mg other regimens (Month 12): number analyzed (Participants) | 5
  5 mg other regimens (Month 12) | 20.6 (500)
  5 mg other regimens (Month 24): number analyzed (Participants) | 3
  5 mg other regimens (Month 24) | 91.1 (236)
  10 mg QD (Month 6): number analyzed (Participants) | 54
  10 mg QD (Month 6) | 126 (161)
  10 mg QD (Month 9): number analyzed (Participants) | 8
  10 mg QD (Month 9) | 51.1 (167)
  10 mg QD (Month 12): number analyzed (Participants) | 48
  10 mg QD (Month 12) | 86.9 (188)
  10 mg QD (Month 24): number analyzed (Participants) | 41
  10 mg QD (Month 24) | 85.6 (152)
  10 mg QD (Month 36): number analyzed (Participants) | 29
  10 mg QD (Month 36) | 79.9 (143)
  10 mg QD (Month 48): number analyzed (Participants) | 20
  10 mg QD (Month 48) | 81.2 (161)
  10 mg QD (Month 60): number analyzed (Participants) | 11
  10 mg QD (Month 60) | 48.6 (323)
  10 mg QOD (Month 12): number analyzed (Participants) | 2
  10 mg QOD (Month 12) | 102 (576)
  10 mg QOD (Month 24): number analyzed (Participants) | 1
  10 mg QOD (Month 24) | 25.5 (NA) — No variation was calculated.
  10 mg QOD (Month 48): number analyzed (Participants) | 1
  10 mg QOD (Month 48) | 9.08 (NA) — No data on OCA concentration was detected.
  10 mg Q2W (Month 6): number analyzed (Participants) | 1
  10 mg Q2W (Month 6) | 538 (NA) — No variation was calculated.
  10 mg Q2W (Month 9): number analyzed (Participants) | 1
  10 mg Q2W (Month 9) | 566 (NA) — No variation was calculated.
  10 mg Q2W (Month 12): number analyzed (Participants) | 2
  10 mg Q2W (Month 12) | 41.7 (45.6)
  10 mg Q2W (Month 24): number analyzed (Participants) | 2
  10 mg Q2W (Month 24) | 62.5 (35.9)
  10 mg Q2W (Month 36): number analyzed (Participants) | 3
  10 mg Q2W (Month 36) | 96.3 (132)
  10 mg Q2W (Month 48): number analyzed (Participants) | 2
  10 mg Q2W (Month 48) | 70.9 (218)
  10 mg Q2W (Month 60): number analyzed (Participants) | 1
  10 mg Q2W (Month 60) | 83.8 (NA) — No variation was calculated.
  10 mg Q3D (Month 12): number analyzed (Participants) | 1
  10 mg Q3D (Month 12) | 0.861 (NA) — No variation was calculated.

38. Secondary Outcome: PK Population: Serial Concentration of OCA By Dose Regimen
Description: In Month 9, blood samples were collected at predose, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4h, 5 h, and 6 h and PK serial concentrations at different dose regimen are reported.
Time Frame: Month 9
Population: The PK Population included all OCA participants who had at least 1 confirmed fasted analyzable sample. Participants fasted for approximately 8 hours prior to the visit and had no major protocol deviations that potentially affected exposure levels.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 13
ng/mL
  5 mg QD (Predose): number analyzed (Participants) | 3
  5 mg QD (Predose) | 61.2 (315)
  5 mg QD (0.5 h): number analyzed (Participants) | 3
  5 mg QD (0.5 h) | 109 (66.1)
  5 mg QD (0.75 h): number analyzed (Participants) | 3
  5 mg QD (0.75 h) | 158 (35.6)
  5 mg QD (1 h): number analyzed (Participants) | 3
  5 mg QD (1 h) | 173 (56.4)
  5 mg QD (1.5 h): number analyzed (Participants) | 3
  5 mg QD (1.5 h) | 137 (53.2)
  5 mg QD (2 h): number analyzed (Participants) | 3
  5 mg QD (2 h) | 100 (100)
  5 mg QD (2.5 h): number analyzed (Participants) | 3
  5 mg QD (2.5 h) | 90.1 (93.0)
  5 mg QD (3 h): number analyzed (Participants) | 3
  5 mg QD (3 h) | 64.7 (47.1)
  5 mg QD (4 h): number analyzed (Participants) | 3
  5 mg QD (4 h) | 71.6 (179)
  5 mg QD (5 h): number analyzed (Participants) | 3
  5 mg QD (5 h) | 193 (150)
  5 mg QD (6 h): number analyzed (Participants) | 3
  5 mg QD (6 h) | 199 (203)
  5 mg QOD (Predose): number analyzed (Participants) | 1
  5 mg QOD (Predose) | 396 (NA) — No variation was calculated.
  5 mg QOD (0.5 h): number analyzed (Participants) | 1
  5 mg QOD (0.5 h) | 236 (NA) — No variation was calculated.
  5 mg QOD (0.75 h): number analyzed (Participants) | 1
  5 mg QOD (0.75 h) | 211 (NA) — No variation was calculated.
  5 mg QOD (1 h): number analyzed (Participants) | 1
  5 mg QOD (1 h) | 217 (NA) — No variation was calculated.
  5 mg QOD (1.5 h): number analyzed (Participants) | 1
  5 mg QOD (1.5 h) | 232 (NA) — No variation was calculated.
  5 mg QOD (2 h): number analyzed (Participants) | 1
  5 mg QOD (2 h) | 243 (NA) — No variation was calculated.
  5 mg QOD (2.5 h): number analyzed (Participants) | 1
  5 mg QOD (2.5 h) | 240 (NA) — No variation was calculated.
  5 mg QOD (3 h): number analyzed (Participants) | 1
  5 mg QOD (3 h) | 171 (NA) — No variation was calculated.
  5 mg QOD (4 h): number analyzed (Participants) | 1
  5 mg QOD (4 h) | 117 (NA) — No variation was calculated.
  5 mg QOD (5 h): number analyzed (Participants) | 1
  5 mg QOD (5 h) | 282 (NA) — No variation was calculated.
  5 mg QOD (6 h): number analyzed (Participants) | 1
  5 mg QOD (6 h) | 544 (NA) — No variation was calculated.
  10 mg QD (Predose): number analyzed (Participants) | 7
  10 mg QD (Predose) | 64.2 (139)
  10 mg QD (0.5 h): number analyzed (Participants) | 6
  10 mg QD (0.5 h) | 142 (55.8)
  10 mg QD (0.75 h): number analyzed (Participants) | 6
  10 mg QD (0.75 h) | 176 (55.5)
  10 mg QD (1 h): number analyzed (Participants) | 6
  10 mg QD (1 h) | 196 (65.5)
  10 mg QD (1.5 h): number analyzed (Participants) | 6
  10 mg QD (1.5 h) | 254 (64.0)
  10 mg QD (2 h): number analyzed (Participants) | 6
  10 mg QD (2 h) | 233 (54.0)
  10 mg QD (2.5 h): number analyzed (Participants) | 6
  10 mg QD (2.5 h) | 206 (80.2)
  10 mg QD (3 h): number analyzed (Participants) | 6
  10 mg QD (3 h) | 217 (90.7)
  10 mg QD (4 h): number analyzed (Participants) | 6
  10 mg QD (4 h) | 151 (74.4)
  10 mg QD (5 h): number analyzed (Participants) | 6
  10 mg QD (5 h) | 180 (80.0)
  10 mg QD (6 h): number analyzed (Participants) | 6
  10 mg QD (6 h) | 214 (77.9)
  10 mg Q2W (Predose): number analyzed (Participants) | 2
  10 mg Q2W (Predose) | 370 (65.8)
  10 mg Q2W (0.5 h): number analyzed (Participants) | 2
  10 mg Q2W (0.5 h) | 490 (52.6)
  10 mg Q2W (P0.75 h): number analyzed (Participants) | 2
  10 mg Q2W (P0.75 h) | 593 (68.2)
  10 mg Q2W (1 h): number analyzed (Participants) | 2
  10 mg Q2W (1 h) | 633 (69.5)
  10 mg Q2W (1.5 h): number analyzed (Participants) | 1
  10 mg Q2W (1.5 h) | 425 (NA) — No variation was calculated.
  10 mg Q2W (2 h): number analyzed (Participants) | 2
  10 mg Q2W (2 h) | 769 (64.5)
  10 mg Q2W (2.5 h): number analyzed (Participants) | 2
  10 mg Q2W (2.5 h) | 716 (75.1)
  10 mg Q2W (3 h): number analyzed (Participants) | 2
  10 mg Q2W (3 h) | 602 (77.2)
  10 mg Q2W (4 h): number analyzed (Participants) | 2
  10 mg Q2W (4 h) | 422 (116)
  10 mg Q2W (5 h): number analyzed (Participants) | 2
  10 mg Q2W (5 h) | 758 (84.4)
  10 mg Q2W (6 h): number analyzed (Participants) | 2
  10 mg Q2W (6 h) | 728 (169)

39. Secondary Outcome: PK Population: Area Under The Concentration-Time Curve (AUC) From 0 to 6 Hours Post-dose (AUC0-6h) Of Participants Who Received 5 mg QD OCA and With CP Score=Non-Cirrhotic (NC)
Description: In Month 9, blood samples were collected at predose, 0.5h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4h, 5 h, and 6 h for PK analysis in participants who received 5 mg QD OCA with CP Score=NC.
Time Frame: Month 9
Population: Participants in the PK population that had the appropriate CP Score, had received the assigned dosage according to the dosage regimen and had an analyzable sample at month 9.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
h*ng/mL | 758 (NA) — No variation was calculated.

40. Secondary Outcome: PK Population: AUC From 0 to 24 Hours Post-dose (AUC0-24h) Of Participants Who Received 5 mg QD OCA and With CP Score=NC
Description: as for outcome 39
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
h*ng/mL | 3710 (NA) — No variation was calculated.

41. Secondary Outcome: PK Population: Maximum Observed Concentration (Cmax) Of Participants Who Received 5mg QD OCA and With CP Score=NC
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 5 mg QD OCA with CP Score=NC.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 317 (NA) — No variation was calculated.

42. Secondary Outcome: PK Population: Time to Cmax (Tmax) Of Participants Who Received 5mg QD OCA and With CP Score=NC
Description: as for outcome 41
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
hours | 6.0 [6.0 to 6.0]

43. Secondary Outcome: PK Population: Metabolite to Parent Ratio of AUC0-6h (MRAUC) Of Participants Who Received 5mg QD OCA and With CP Score=NC
Description: as for outcome 41
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ratio | 15.9 (NA) — No variation was calculated.

44. Secondary Outcome: PK Population: Metabolite to Parent Ratio of Cmax (MRCmax) Of Participants Who Received 5mg QD OCA and With CP Score=NC
Description: as for outcome 41
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ratio | 8.93 (NA) — No variation was calculated.

45. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 5 mg QD OCA and With CP Score=A
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 5 mg QD OCA with CP Score=A.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
h*ng/mL | 889 (133)

46. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 5 mg QD OCA and With CP Score=A
Description: as for outcome 45
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
h*ng/mL | 4040 (129)

47. Secondary Outcome: PK Population: Cmax Of Participants Who Received 5mg QD OCA and With CP Score=A
Description: as for outcome 45
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ng/mL | 275 (117)

48. Secondary Outcome: PK Population: Tmax Of Participants Who Received 5mg QD OCA and With CP Score=A
Description: as for outcome 45
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
hours | 3.38 [0.750 to 6.0]

49. Secondary Outcome: PK Population: Concentration at 24 Hours Post-dose (Ctrough) Of Participants Who Received 5mg QD OCA and With CP Score=A
Description: as for outcome 45
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ng/mL | 149 (22.2)

50. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 5mg QD OCA and With CP Score=A
Description: as for outcome 45
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ratio | 8.41 (50.8)

51. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 5mg QD OCA and With CP Score=A
Description: as for outcome 45
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ratio | 3.77 (64.5)

52. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 5mg QD OCA and With CP Score=B
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 5 mg QD OCA with CP Score=B.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 242 (NA) — No variation was calculated.

53. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 5 mg QOD OCA and With CP Score=NC
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 5 mg QOD OCA with CP Score=NC.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
h*ng/mL | 1480 (NA) — No variation was calculated.

54. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 5 mg QOD OCA and With CP Score=NC
Description: as for outcome 53
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
h*ng/mL | 9940 (NA) — No variation was calculated.

55. Secondary Outcome: PK Population: Cmax Of Participants Who Received 5mg QOD OCA and With CP Score=NC
Description: as for outcome 53
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 544 (NA) — No variation was calculated.

56. Secondary Outcome: PK Population: Tmax Of Participants Who Received 5mg QOD OCA and With CP Score=NC
Description: as for outcome 53
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
hours | 6.0 [6.0 to 6.0]

57. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 5mg QOD OCA and With CP Score=NC
Description: as for outcome 53
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 396 (NA) — No variation was calculated.

58. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 5mg QOD OCA and With CP Score=NC
Description: as for outcome 53
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ratio | 26.6 (NA) — No variation was calculated.

59. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 5mg QOD OCA and With CP Score=NC
Description: as for outcome 53
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ratio | 15.8 (NA) — No variation was calculated.

60. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 10 mg QD OCA and With CP Score=NC
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 10 mg QOD OCA with CP Score=NC.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
h*ng/mL | 1090 (98.4)

61. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 10 mg QD OCA and With CP Score=NC
Description: as for outcome 60
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
h*ng/mL | 3820 (91.7)

62. Secondary Outcome: PK Population: Cmax Of Participants Who Received 10 mg QD OCA and With CP Score=NC
Description: as for outcome 60
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ng/mL | 289 (74.5)

63. Secondary Outcome: PK Population: Tmax Of Participants Who Received 10 mg QD OCA and With CP Score=NC
Description: as for outcome 60
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
hours | 1.50 [1.50 to 3.00]

64. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 10 mg QD OCA and With CP Score=NC
Description: as for outcome 60
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 4
ng/mL | 50.6 (148)

65. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 10 mg QD OCA and With CP Score=NC
Description: as for outcome 60
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ratio | 13.8 (151)

66. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 10 mg QD OCA and With CP Score=NC
Description: as for outcome 60
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ratio | 4.02 (107)

67. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 10 mg QD OCA and With CP Score=A
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 10 mg QD OCA with CP Score=A.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
h*ng/mL | 1310 (11.9)

68. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 10 mg QD OCA and With CPS Score=A
Description: as for outcome 67
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
h*ng/mL | 4280 (26.1)

69. Secondary Outcome: PK Population: Cmax Of Participants Who Received 10 mg QD OCA and With CP Score=A
Description: as for outcome 67
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ng/mL | 334 (6.71)

70. Secondary Outcome: PK Population: Tmax Of Participants Who Received 10 mg QD OCA and With CPS Score=A
Description: as for outcome 67
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
hours | 1.50 [0.750 to 2.50]

71. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 10 mg QD OCA and With CP Score=A
Description: as for outcome 67
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ng/mL | 55.2 (414)

72. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 10 mg QD OCA and With CP Score=A
Description: as for outcome 67
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ratio | 2.94 (15.5)

73. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 10 mg QD OCA and With CP Score=A
Description: as for outcome 67
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ratio | 1.48 (21.8)

74. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 10 mg Q2W OCA and With CP Score=B
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 10 mg Q2W OCA with CP Score=B.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
h*ng/mL | 3770 (84.9)

75. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 10 mg Q2W OCA and With CP Score=B
Description: as for outcome 74
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
h*ng/mL | 13900 (113)

76. Secondary Outcome: PK Population: Cmax Of Participants Who Received 10 mg Q2W OCA and With CP Score=B
Description: as for outcome 74
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ng/mL | 916 (101)

77. Secondary Outcome: PK Population: Tmax Of Participants Who Received 10 mg Q2W OCA and With CP Score=B
Description: as for outcome 74
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
hours | 4.0 [2.0 to 6.0]

78. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 10 mg Q2W OCA and With CP Score=B
Description: as for outcome 74
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 566 (NA) — No variation was calculated.

79. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 10 mg Q2W OCA and With CP Score=B
Description: as for outcome 74
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ratio | 12.6 (450)

80. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 10 mg Q2W OCA and With CP Score=B
Description: as for outcome 74
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ratio | 7.13 (315)

81. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 5 mg QD OCA and With MELD Category=A
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 5 mg QD OCA with MELD Category=A.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
h*ng/mL | 1170 (68.0)

82. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 5 mg QD OCA and With MELD Category=A
Description: as for outcome 81
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
h*ng/mL | 5490 (60.2)

83. Secondary Outcome: PK Population: Cmax Of Participants Who Received 5 mg QD OCA and With MELD Category=A
Description: as for outcome 81
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ng/mL | 410 (37.4)

84. Secondary Outcome: PK Population: Tmax Of Participants Who Received 5 mg QD OCA and With MELD Category=A
Description: as for outcome 81
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
hours | 6.0 [6.0 to 6.0]

85. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 5 mg QD OCA and With MELD Category=A
Description: as for outcome 81
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 174 (NA) — No variation was calculated.

86. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 5 mg QD OCA and With MELD Category=A
Description: as for outcome 81
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ratio | 13.7 (21.1)

87. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 5 mg QD OCA and With MELD Category=A
Description: as for outcome 81
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ratio | 7.15 (32.3)

88. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 5 mg QD OCA and With MELD Category=B
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 5 mg QD OCA with MELD Category=B.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
h*ng/mL | 436 (NA) — No variation was calculated.

89. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 5 mg QD OCA and With MELD Category=B
Description: as for outcome 88
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
h*ng/mL | 2000 (NA) — No variation was calculated.

90. Secondary Outcome: PK Population: Cmax Of Participants Who Received 5 mg QD OCA and With MELD Category=B
Description: as for outcome 88
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 143 (NA) — No variation was calculated.

91. Secondary Outcome: PK Population: Tmax Of Participants Who Received 5 mg QD OCA and With MELD Category=B
Description: as for outcome 88
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
hours | 0.750 [0.750 to 0.750]

92. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 5 mg QD OCA and With MELD Category=B
Description: as for outcome 88
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ng/mL | 176 (47.9)

93. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 5 mg QD OCA and With MELD Category=B
Description: as for outcome 88
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ratio | 5.99 (NA) — No variation was calculated.

94. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 5 mg QD OCA and With MELD Category=B
Description: as for outcome 88
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ratio | 2.48 (NA) — No variation was calculated.

95. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 5 mg QOD OCA and With MELD Category=A
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 5 mg QOD OCA with MELD Category=A.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
h*ng/mL | 1480 (NA) — No variation was calculated.

96. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 5 mg QOD OCA and With MELD Category=A
Description: as for outcome 95
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
h*ng/mL | 9940 (NA) — No variation was calculated.

97. Secondary Outcome: PK Population: Cmax Of Participants Who Received 5 mg QOD OCA and With MELD Category=A
Description: as for outcome 95
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 544 (NA) — No variation was calculated.

98. Secondary Outcome: PK Population: Tmax Of Participants Who Received 5 mg QOD OCA and With MELD Category=A
Description: as for outcome 95
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
hours | 6.0 [6.0 to 6.0]

99. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 5 mg QOD OCA and With MELD Category=A
Description: as for outcome 95
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 396 (NA) — No variation was calculated.

100. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 5 mg QOD OCA and With MELD Category=A
Description: as for outcome 95
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ratio | 26.6 (NA) — No variation was calculated.

101. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 5 mg QOD OCA and With MELD Category=A
Description: as for outcome 95
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ratio | 15.8 (NA) — No variation was calculated.

102. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 10 mg QD OCA and With MELD Category=A
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 10 mg QD OCA with MELD Category=A.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
h*ng/mL | 886 (55.6)

103. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 10 mg QD OCA and With MELD Category=A
Description: as for outcome 102
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
h*ng/mL | 2860 (35.5)

104. Secondary Outcome: PK Population: Cmax Of Participants Who Received 10 mg QD OCA and With MELD Category=A
Description: as for outcome 102
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ng/mL | 240 (35.1)

105. Secondary Outcome: PK Population: Tmax Of Participants Who Received 10 mg QD OCA and With MELD Category=A
Description: as for outcome 102
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
hours | 1.50 [1.50 to 3.00]

106. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 10 mg QD OCA and With MELD Category=A
Description: as for outcome 102
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 4
ng/mL | 25.8 (188)

107. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 10 mg QD OCA and With MELD Category=A
Description: as for outcome 102
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ratio | 6.04 (162)

108. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 10 mg QD OCA and With MELD Category=A
Description: as for outcome 102
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ratio | 1.92 (50.6)

109. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 10 mg QD OCA and With MELD Category=B
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 10 mg QD OCA with MELD Category=B.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
h*ng/mL | 1610 (44.6)

110. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 10 mg QD OCA and With MELD Category=B
Description: as for outcome 109
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
h*ng/mL | 5700 (48.7)

111. Secondary Outcome: PK Population: Cmax Of Participants Who Received 10 mg QD OCA and With MELD Category=B
Description: as for outcome 109
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ng/mL | 403 (39.4)

112. Secondary Outcome: PK Population: Tmax Of Participants Who Received 10 mg QD OCA and With MELD Category=B
Description: as for outcome 109
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
hours | 1.50 [0.750 to 2.50]

113. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 10 mg QD OCA and With MELD Category=B
Description: as for outcome 109
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ng/mL | 136 (14.9)

114. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 10 mg QD OCA and With MELD Category=B
Description: as for outcome 109
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ratio | 6.73 (212)

115. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 10 mg QD OCA and With MELD Category=B
Description: as for outcome 109
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ratio | 3.11 (147)

116. Secondary Outcome: PK Population: AUC0-6h Of Participants Who Received 10 mg Q2W OCA and With MELD Category=B
Description: In Month 9, blood samples were collected at predose to 6 h for PK analysis in participants who received 10 mg Q2W OCA with MELD Category=B.
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
h*ng/mL | 3770 (84.9)

117. Secondary Outcome: PK Population: AUC0-24h Of Participants Who Received 10 mg Q2W OCA and With MELD Category=B
Description: as for outcome 116
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
h*ng/mL | 13900 (113)

118. Secondary Outcome: PK Population: Cmax Of Participants Who Received 10 mg Q2W OCA and With MELD Category=B
Description: as for outcome 116
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ng/mL | 916 (101)

119. Secondary Outcome: PK Population: Tmax Of Participants Who Received 10 mg Q2W OCA and With MELD Category=B
Description: as for outcome 116
Time Frame: Month 9
Population: as for outcome 39
Measure: Median (Full Range); unit: hours
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
hours | 4.0 [2.0 to 6.0]

120. Secondary Outcome: PK Population: Ctrough Of Participants Who Received 10 mg Q2W OCA and With MELD Category=B
Description: as for outcome 116
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 566 (NA) — No variation was calculated.

121. Secondary Outcome: PK Population: MRAUC Of Participants Who Received 10 mg Q2W OCA and With MELD Category=B
Description: as for outcome 116
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ratio | 12.6 (450)

122. Secondary Outcome: PK Population: MRCmax Of Participants Who Received 10 mg Q2W OCA and With MELD Category=B
Description: as for outcome 116
Time Frame: Month 9
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ratio | 7.13 (315)

123. Secondary Outcome: PK Population: Trough Concentrations Of Cirrhotic Participants Who Received 5 mg QD OCA
Description: The trough concentration of OCA in the cirrhotic participants who received 5 mg QD OCA was reported.
Time Frame: Months 3, 6, 12, 24, and 48
Population: Participants in the PK population that had data available for cirrhosis status, mean trough concentrations by presence or absence of cirrhosis and dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 13
ng/mL
  Month 3: number analyzed (Participants) | 1
  Month 3 | 295 (NA) — No variation was calculated.
  Month 6: number analyzed (Participants) | 3
  Month 6 | 291 (166)
  Month 12: number analyzed (Participants) | 10
  Month 12 | 227 (127)
  Month 24: number analyzed (Participants) | 1
  Month 24 | 127 (NA) — No variation was calculated.
  Month 48: number analyzed (Participants) | 1
  Month 48 | 849 (NA) — No variation was calculated.

124. Secondary Outcome: PK Population: Trough Concentrations Of Non-Cirrhotic Participants Who Received 5 mg QD OCA
Description: The trough concentration of OCA in the non-cirrhotic participants who received 5 mg QD OCA was reported.
Time Frame: Months 3, 6, 9, 12, and 24
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 23
ng/mL
  Month 3: number analyzed (Participants) | 12
  Month 3 | 77.4 (157)
  Month 6: number analyzed (Participants) | 10
  Month 6 | 55.9 (85.1)
  Month 9: number analyzed (Participants) | 1
  Month 9 | 127 (NA) — No variation was calculated.
  Month 12: number analyzed (Participants) | 7
  Month 12 | 96.0 (94.7)
  Month 24: number analyzed (Participants) | 2
  Month 24 | 45.4 (693)

125. Secondary Outcome: PK Population: Trough Concentrations Of Cirrhotic Participants Who Received 5 mg QOD OCA
Description: The trough concentration of OCA in the cirrhotic participants who received 5 mg QOD OCA was reported.
Time Frame: Months 6, 12, and 24
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 5
ng/mL
  Month 6: number analyzed (Participants) | 1
  Month 6 | 1050 (NA) — No variation was calculated.
  Month 12: number analyzed (Participants) | 1
  Month 12 | 48.0 (NA) — No variation was calculated.
  Month 24: number analyzed (Participants) | 3
  Month 24 | 134 (17.1)

126. Secondary Outcome: PK Population: Trough Concentrations Of Non-Cirrhotic Participants Who Received 5 mg QOD OCA
Description: The trough concentration of OCA in the non-cirrhotic participants who received 5 mg QOD OCA was reported.
Time Frame: Months 3, 6, and 12
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 4
ng/mL
  Month 3: number analyzed (Participants) | 2
  Month 3 | 97.2 (53.9)
  Month 6: number analyzed (Participants) | 1
  Month 6 | 85.4 (NA) — No variation was calculated.
  Month 12: number analyzed (Participants) | 2
  Month 12 | 200 (184)

127. Secondary Outcome: PK Population: Trough Concentrations Of Cirrhotic Participants Who Received 5 mg QW OCA
Description: The trough concentration of OCA in the cirrhotic participants who received 5 mg QW OCA was reported.
Time Frame: Months 6 and 12
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 4
ng/mL
  Month 6: number analyzed (Participants) | 1
  Month 6 | 56.7 (NA) — No variation was calculated.
  Month 12: number analyzed (Participants) | 3
  Month 12 | 116 (395)

128. Secondary Outcome: PK Population: Trough Concentrations Of Non-Cirrhotic Participants Who Received 5 mg QW OCA
Description: In Month 12, the trough concentration of OCA in the non-cirrhotic participants who received 5 QW QOD OCA was reported.
Time Frame: Month 12
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 179 (NA) — No variation was calculated.

129. Secondary Outcome: PK Population: Trough Concentrations Of Cirrhotic Participants Who Received 5 mg Q2W OCA
Description: The trough concentration of OCA in the cirrhotic participants who received 5 mg Q2W OCA was reported.
Time Frame: Months 6, 24, 36 and 48
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 3
ng/mL
  Month 6: number analyzed (Participants) | 1
  Month 6 | 131 (NA) — No variation was calculated.
  Month 24: number analyzed (Participants) | 1
  Month 24 | 497 (NA) — No variation was calculated.
  Month 36: number analyzed (Participants) | 1
  Month 36 | 117 (NA) — No variation was calculated.
  Month 48: number analyzed (Participants) | 1
  Month 48 | 271 (NA) — No variation was calculated.

130. Secondary Outcome: PK Population: Trough Concentrations Of Non-Cirrhotic Participants Who Received 5 mg Q2W OCA
Description: The trough concentration of OCA in the non-cirrhotic participants who received 5 Q2W QOD OCA was reported.
Time Frame: Months 3, 6, 12, 24, 36, and 48
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 2
ng/mL
  Month 3: number analyzed (Participants) | 1
  Month 3 | 86.0 (NA) — No variation was calculated.
  Month 6: number analyzed (Participants) | 1
  Month 6 | 122 (NA) — No variation was calculated.
  Month 12: number analyzed (Participants) | 1
  Month 12 | 250 (NA) — No variation was calculated.
  Month 24: number analyzed (Participants) | 1
  Month 24 | 497 (NA) — No variation was calculated.
  Month 36: number analyzed (Participants) | 1
  Month 36 | 117 (NA) — No variation was calculated.
  Month 48: number analyzed (Participants) | 1
  Month 48 | 271 (NA) — No variation was calculated.

131. Secondary Outcome: PK Population: Trough Concentrations Of Cirrhotic Participants Who Received 10 mg QD OCA
Description: The trough concentration of OCA in the cirrhotic participants who received 10 mg QD OCA was reported.
Time Frame: Months 6, 9, 12, 24, 36, and 60
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 11
ng/mL
  Month 6: number analyzed (Participants) | 2
  Month 6 | 142 (242)
  Month 9: number analyzed (Participants) | 1
  Month 9 | 7.74 (NA) — No variation was calculated.
  Month 12: number analyzed (Participants) | 8
  Month 12 | 133 (489)
  Month 24: number analyzed (Participants) | 2
  Month 24 | 396 (61.7)
  Month 36: number analyzed (Participants) | 1
  Month 36 | 346 (NA) — No variation was calculated.
  Month 60: number analyzed (Participants) | 1
  Month 60 | 290 (NA) — No variation was calculated.

132. Secondary Outcome: PK Population: Trough Concentrations Of Non-Cirrhotic Participants Who Received 10 mg QD OCA
Description: The trough concentration of OCA in the non-cirrhotic participants who received 10 QD QOD OCA was reported.
Time Frame: Months 6, 9, 12, 24, and 36
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 21
ng/mL
  Month 6: number analyzed (Participants) | 7
  Month 6 | 127 (601)
  Month 9: number analyzed (Participants) | 2
  Month 9 | 74.5 (10.6)
  Month 12: number analyzed (Participants) | 8
  Month 12 | 73.3 (102)
  Month 24: number analyzed (Participants) | 9
  Month 24 | 100 (216)
  Month 36: number analyzed (Participants) | 2
  Month 36 | 98.5 (1730)

133. Secondary Outcome: PK Population: Trough Concentrations Of Cirrhotic Participants Who Received 10 mg QOD OCA
Time Frame: Months 3, 6, 9, 12, 24, 36, 48, and 60
Population: No participant was tested for this outcome measure.
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 0

134. Secondary Outcome: PK Population: Trough Concentrations Of Non-Cirrhotic Participants Who Received 10 mg QOD OCA
Description: In Month 12, the trough concentration of OCA in the non-cirrhotic participants who received 10 mg QOD OCA was reported.
Time Frame: Month 12
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 26.9 (NA) — No variation was calculated.

135. Secondary Outcome: PK Population: Trough Concentrations Of Cirrhotic Participants Who Received 10 mg Q2W OCA
Description: In Month 6, the trough concentration of OCA in the cirrhotic participants who received 10 mg Q2W OCA was reported.
Time Frame: Month 6
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 538 (NA) — No variation was calculated.

136. Secondary Outcome: PK Population: Trough Concentrations Of Non-Cirrhotic Participants Who Received 10 mg Q2W OCA
Description: In Month 6, the trough concentration of OCA in the non-cirrhotic participants who received 10 mg Q2W OCA was reported.
Time Frame: Month 6
Population: as for outcome 123
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 1
ng/mL | 566 (NA) — No variation was calculated.

ADVERSE EVENTS:
Time Frame: Baseline up to the last IP dose plus 30 days and prior to commercial OCA initiation date, approximately 7 years
Arm/Group | Obeticholic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 16/168 | 12/166
Serious Adverse Events (participants affected / at risk) | 53/168 | 53/166
Other Adverse Events (participants affected / at risk) | 156/168 | 146/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obeticholic Acid (N=168) | Placebo (N=166)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 | 5
Ascites (Gastrointestinal disorders) | 2 | 4
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 1
Corynebacterium bacteraemia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Spinal cord abscess (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Viral pericarditis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 2
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 1
Jaundice hepatocellular (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 3 | 5
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Demyelination (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Disease progression (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 2 | 1
Chest discomfort (General disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1
Tumour marker increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Oesophageal variceal ligation (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obeticholic Acid (N=168) | Placebo (N=166)
Pruritus (Skin and subcutaneous tissue disorders) | 131 | 85
Rash (Skin and subcutaneous tissue disorders) | 10 | 6
Abdominal pain upper (Gastrointestinal disorders) | 25 | 12
Nausea (Gastrointestinal disorders) | 25 | 21
Abdominal pain (Gastrointestinal disorders) | 21 | 17
Diarrhoea (Gastrointestinal disorders) | 21 | 26
Varices oesophageal (Gastrointestinal disorders) | 20 | 27
Constipation (Gastrointestinal disorders) | 19 | 10
Ascites (Gastrointestinal disorders) | 18 | 20
Abdominal distension (Gastrointestinal disorders) | 15 | 8
Portal hypertensive gastropathy (Gastrointestinal disorders) | 14 | 7
Vomiting (Gastrointestinal disorders) | 14 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 6
Dyspepsia (Gastrointestinal disorders) | 9 | 8
Oedema peripheral (General disorders) | 31 | 18
Fatigue (General disorders) | 18 | 25
Pyrexia (General disorders) | 12 | 8
Urinary tract infection (Infections and infestations) | 20 | 30
Nasopharyngitis (Infections and infestations) | 18 | 14
Upper respiratory tract infection (Infections and infestations) | 14 | 10
Sinusitis (Infections and infestations) | 11 | 9
Bronchitis (Infections and infestations) | 10 | 8
Influenza (Infections and infestations) | 9 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7
Osteoporosis (Musculoskeletal and connective tissue disorders) | 5 | 11
Headache (Nervous system disorders) | 23 | 21
Dizziness (Nervous system disorders) | 10 | 14
Hepatic encephalopathy (Nervous system disorders) | 7 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 9 | 8
Jaundice (Hepatobiliary disorders) | 8 | 10
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 11
Blood bilirubin increased (Investigations) | 19 | 25
Anaemia (Blood and lymphatic system disorders) | 10 | 13
Splenomegaly (Blood and lymphatic system disorders) | 3 | 9
Insomnia (Psychiatric disorders) | 12 | 16
Hypertension (Vascular disorders) | 9 | 7

LIMITATIONS AND CAVEATS:
The estimated effect of treatment from the ITT population was underpowered and potentially biased, resulting in difficulties in the interpretation of the tests of hypotheses for the primary and key secondary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators must wait 18 months after the study ends to publish their results and a multi-center publication must come first. The sponsor has a 45-day review period with the option to extend it to an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT02308111/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT02308111/SAP_001.pdf